CLINICAL TRIAL: NCT06698484
Title: A Phase II Open Label Single-arm Study to Evaluate Safety and Efficacy of Autologous CD19 CAR-T Cells in Patients With Relapsed/Refractory B- Non-Hodgkin Lymphoma
Brief Title: To Evaluate Safety and Efficacy of Autologous CD19 Chimeric Antigen Receptor (CAR)-T Cells in Relapsed/Refractory B- Non-Hodgkin Lymphoma (B-NHL)
Acronym: CAR-T for NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Plutonet Sdn Bhd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T NHL PTS Plutonet 2021; JEP-2021-224 (Other: Research Ethics Committee Universiti Kebangsaan Malaysia (REC UKM))
Record Dates: First submitted 2024-11-10; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Relapsed/Refractory B- Cell Non-Hodgkin Lymphoma
Keywords: RR B- NHL; CD19 CAR-T cells; malaysia
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient will infuse with autologous CD19 CAR-T cells (Experimental): CD19 CAR-T cells
  Interventions: Drug: CAR-T cells

INTERVENTIONS:
Drug: CAR-T cells — 2×10^6 CAR T cells/kg

SUMMARY:
A Phase II Open-Label Single-arm Study to Evaluate Safety and Efficacy of locally manufactured autologous CD19-directed CAR T-cells in Patients with Relapsed/Refractory B- Non-Hodgkin Lymphoma (B-NHL) or patients not eligible for hematopoietic stem cell transplantation (HCT)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosed with CD19 positive B cell NHL in accordance with WHO classification
* Patients who are refractory to second-line treatment or patients who relapsed after first-line treatment with no available curative options such as autologous or allogeneic haematopoietic stem cell transplantation (HSCT) or relapse within one year of autologous HSCT
* At least one measurable lesion according to revised IWG response criteria
* Age between ≥13to ≤75 years
* Adequate organ function as defined by a creatinine clearance >40 ml/min, serum alanine transaminase (ALT) < 5 times the normal value, serum bilirubin < 3 times the normal value, left ventricular ejection fraction> 45%
* Absolute neutrophil count ≥ 1500/μl, haemoglobin level ≥ 7 g/dl, platelets ≥ 50000/μl.
* Life expectancy >12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Female of childbearing age must have a negative pregnancy test and is on two effective contraception methods
* Male patients must use two effective contraception methods

Exclusion Criteria:

* Active central nervous system (CNS) lymphoma (detected by Imaging study or cerebrospinal fluid (CSF) analysis)
* Active cancer(other than NHL) or receiving cancer treatment
* Evidence of severe lung, heart (New York Heart Association class III/IV, arrhythmia, heart block, uncontrolled hypertension), liver, or renal failure or severe neurologic disorder
* Presence of active autoimmune disease requiring immunosuppressive therapy
* Human Immunodeficiency Virus (HIV) positivity
* Active Hepatitis B, and Hepatitis C infection
* Uncontrolled infection
* Pregnant/nursing female.
* Receiving autologous or allogeneic stem cell transplant within 12 weeks of enrolment

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From day 30, then 3 monthly until 24 months after infusion of CAR-T cells
  The ORR is the sum of patients achieving complete response (CR) and partial response (PR) at day 30, then 3 monthly up to 24 months after receiving CAR T-cells determined by the investigator following Lugano criteria in non-Hodgkin Lymphoma (NHL).
  Response assessment will be determined using a PET CT scan, or other relevant imaging studies and compared to the baseline (pre-CAR-T infusion) study.

SECONDARY OUTCOMES:
overall survival | OS at day 30, 6 months and one year, and 2 years following CAR-T cells infusion
  Overall survival (OS) is defined as the time from the date of CAR-T cell infusion to the date of death from any cause. Patients who are still alive will be censored at the date of last contact.
Incidence of adverse events | From the time of infusion up to 24 months after infusion of CAR-T cells
  Cumulative incidence of CAR-T cell treatment-related adverse events (AEs) graded by ASCT consensus grading criteria for cytokine release syndrome (CRS) and Immune Effector cell-associated Neurotoxicity Syndrome (ICANS) and by common terminology criteria adverse events (CTCAE) versions 5.0 for other AEs in p[articular hematotoxicity and infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No